CLINICAL TRIAL: NCT02032407
Title: A Study of Dapsone Gel in Females With Skin of Color and Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMA-ACZ-13-001
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dapsone Gel (Experimental): Dapsone Gel (Aczone®) applied twice daily to the face for 12 weeks.
  Interventions: Drug: Dapsone Gel

INTERVENTIONS:
Drug: Dapsone Gel — Dapsone Gel (Aczone®) applied twice daily to the face for 12 weeks.
  Other Names: Aczone®

SUMMARY:
This study will evaluate the effect of dapsone gel in female subjects with skin of color (Fitzpatrick Skin Types IV, V, and VI) with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acne vulgaris
* Medium to dark complexion (Fitzpatrick Skin Type IV, V or VI)
* Willing to avoid excessive or prolonged exposure of the face to ultraviolet light (eg, sunlight, tanning beds) throughout the study

Exclusion Criteria:

* Received treatment with botulinum toxin of any serotype in the face within 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapsone Gel
Started | 68
Completed | 63
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Pregnancy | 1
Not completed — Other Miscellaneous Reasons | 2

BASELINE CHARACTERISTICS:
Population: Modified Intent-to treat population included all enrolled participants who received at least one application of study treatment and had at least one post-Baseline efficacy assessment.
Arm/Group | Dapsone Gel
Number analyzed (Participants) | 67
Age, Customized [Number; unit: participants]
  18 to <30 years | 32
  ≥30 to <50 years | 32
  ≥50 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Global Assessment of Acne Severity (GAAS) Score by Physician
Description: The investigator evaluated the participant's acne severity using the 5-point GAAS grading scale: 0= No evidence of facial acne vulgaris to 4= Significant degree of inflammatory disease; papules/pustules were a predominant feature; a few nodulo-cystic lesions could have been present; comedones (small pumps on the skin caused by acne) could have been present. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: Modified Intent-to treat (mITT) population included all enrolled participants who received at least one application of study treatment and had at least one post-Baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dapsone Gel
Number analyzed (Participants) | 67
score on a scale
  Baseline | 2.8 (0.72)
  Change from Baseline at Week 12 | -1.2 (0.88)

2. Secondary Outcome: Change From Baseline in the GAAS
Description: as for outcome 1
Time Frame: Baseline, Weeks 2 and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dapsone Gel
Number analyzed (Participants) | 67
score on a scale
  Baseline | 2.8 (0.72)
  Change from Baseline at Week 2 | -0.3 (0.63)
  Change from Baseline at Week 6 | -0.6 (0.74)

3. Secondary Outcome: Percent Change From Baseline in Total Lesion Counts
Description: The investigator evaluated Inflammatory (papule, pustule and nodule/cyst) and Non-inflammatory (blackhead and whitehead) lesions. A papule is a small, red, solid elevation less than 1.0 cm in diameter, a pustule is a small, circumscribed elevation of the skin that contains yellow-white exudate and a nodule/cyst is a circumscribed, elevated, solid lesion generally more than 0.5 cm in diameter with palpable depth. The total lesion count was the sum of the inflammatory and non-inflammatory lesion counts. A negative percent change from baseline indicates a reduction in lesion counts (improvement).
Time Frame: Baseline, Weeks 2, 6 and 12
Population: Participants from the Modified Intent-to treat (mITT) population, all enrolled participants who received at least one application of study treatment and had at least one post-Baseline efficacy assessment, with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dapsone Gel
Number analyzed (Participants) | 67
percent change
  Change from Baseline at Week 2 | -16.0 (23.45)
  Change from Baseline at Week 6 (n=61) | -30.0 (26.15)
  Change from Baseline at Week 12 (n=63) | -52.0 (26.96)

4. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Counts
Description: The investigator evaluated Inflammatory lesions (papule, pustule and nodule/cyst). A negative percent change from baseline indicates a reduction in lesion counts (improvement).
Time Frame: Baseline, Weeks 2, 6 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dapsone Gel
Number analyzed (Participants) | 67
percent change
  Change from Baseline at Week 2 | -25.0 (32.01)
  Change from Baseline at Week 6 (n=61) | -48.0 (26.72)
  Change from Baseline at Week 12 (n=63) | -65.0 (23.31)

5. Secondary Outcome: Percent Change From Baseline in Non-Inflammatory Lesion Counts
Description: The investigator evaluated Non-inflammatory (blackhead and whitehead) lesions. A negative percent change from baseline indicates a reduction in lesion counts (improvement).
Time Frame: Baseline, Weeks 2, 6 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dapsone Gel
Number analyzed (Participants) | 67
percent change
  Change from Baseline at Week 2 | -9.8 (32.03)
  Change from Baseline at Week 6 (n=61) | -16.0 (36.19)
  Change from Baseline at Week 12 (n=63) | -41.0 (34.15)

6. Secondary Outcome: Percentage of Participants With 0 (None) or 1 (Minimal) on the GAAS
Description: The investigator evaluated the participant's acne severity using the 5-point GAAS grading scale: 0= No evidence of facial acne vulgaris to 4= Significant degree of inflammatory disease; papules/pustules were a predominant feature; a few nodulo-cystic lesions could have been present; comedones (small pumps on the skin caused by acne) could have been present. The percentage of participants with a score of 0=none or 1=minimal is reported.
Time Frame: Weeks 2, 6 and 12
Population: Participants from the mITT, all enrolled participants who received at least one application of study treatment and had at least one post-Baseline efficacy assessment, with data available at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Dapsone Gel
Number analyzed (Participants) | 67
percentage of participants
  Week 2 | 6.0
  Week 6 (n=61) | 13.1
  Week 12 (n=63) | 42.9

7. Secondary Outcome: Acne Symptom and Impact Scale (ASIS) Sign Domain Score
Description: The participant assessed signs of acne vulgaris using the ASIS. The sign domain is a composite of 9 items of the 17 items on the overall scale. Each of the items is answered on a 5-point scale: 0 (best) to 4 (worst). The sign domain score is calculated as the average of the 9 items for a total possible score of 0 to 4. Higher scores indicate the presence of more severe signs of acne.
Time Frame: Weeks 2, 6 and 12
Population: Participants from the mITT population, all enrolled participants who received at least one application of study treatment and had at least one post-Baseline efficacy assessment, with data at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dapsone Gel
Number analyzed (Participants) | 67
score on a scale
  Week 2 | 1.7 (0.72)
  Week 6 (n=60) | 1.3 (0.68)
  Week 12 (n=63) | 1.1 (0.67)

8. Secondary Outcome: ASIS Impact Domain Score
Description: The participant assessed the impact of acne vulgaris using the ASIS. The impact domain is a composite of 8 items assessing the psychosocial impacts (6 items emotional and 2 items social) of the 17 items on the overall scale. Each of the items is answered on a 5-point scale: 0 (best) to 4 (worst). The impact domain score is calculated as the average of the 8 items for a total possible score of 0 to 4. Higher scores on the ASIS Impact Domain indicate greater negative impact of acne on health-related quality of life and appearance.
Time Frame: Weeks 2, 6 and 12
Population: Participants from the mITT population, all enrolled participants who received at least one application of study treatment and had at least one post-Baseline efficacy assessment, with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dapsone Gel
Number analyzed (Participants) | 67
score on a scale
  Week 2 | 1.6 (0.91)
  Week 6 (n=60) | 1.3 (0.91)
  Week 12 (n=63) | 1.1 (0.91)

ADVERSE EVENTS:
Arm/Group | Dapsone Gel
Serious Adverse Events (participants affected / at risk) | 1/68
Other Adverse Events (participants affected / at risk) | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapsone Gel (N=68)
Spontaneous abortion (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.